CLINICAL TRIAL: NCT06561438
Title: Postoperative Pain Management Following Laparoscopic Cholecystectomy- Vortioxetine
Brief Title: Postoperative Pain Management Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hoda Mohamed, Principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/2024
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
Keywords: laparoscopic; 5-HT3 and 5-HT7 receptors inhibition; post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The patient will not be administered with any drug/placebo before the surgery
- Intervention arm (Experimental): 20 mg oral vortioxetine tablet 2 hours before the procedure
  Interventions: Drug: Vortioxetine 20Mg Tab

INTERVENTIONS:
Drug: Vortioxetine 20Mg Tab — 20 mg oral vortioxetine tablet 2 hours before the procedure
  Arms: Intervention arm

SUMMARY:
Postoperative pain management is essential and the inability to treat acute pain appropriately in the first 48 postoperative hours represents a risk factor for developing chronic pain. No. study has investigated Vortioxetine as an adjuvant to standard care for postoperative pain management in patients undergoing LC

DETAILED DESCRIPTION:
Postoperative pain is a main challenge for delayed hospital discharge in Laparoscopic cholecystectomy. . Postoperative pain management is essential and the inability to treat acute pain appropriately in the first 48 postoperative hours represents a risk factor for developing chronic pain. Vortioxetine (VO) is a multimodal serotonergic antidepressant with a unique mechanism of action that is effective in treating neuropathic pain. The purpose of this study is evaluating the efficacy and tolerability of preoperative oral administration of Vortioxetine on postoperative pain control in patients undergoing LC

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo elective LC.
* Adults (males and/or females) between the ages of 18-70 years old.

Exclusion Criteria:

* Chronic pain other than cholelithiasis.
* Patients who received analgesics or sedatives 24 h before scheduled surgery.
* Severe hepatic (Child Pugh Class B and C) and renal dysfunction (CrCl <30ml/min)
* Previous allergic response to vortioxetine.
* Pregnancy and lactation
* Patients with communication problems, cognitive dysfunction, or psychological disorders
* Daily corticosteroid use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
VAS score (Visual analogue scale) | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours
  Pain intensity: VAS score from 0 to 100 mm In which 0 means no pain, and 100 means the worst pain possible

SECONDARY OUTCOMES:
Time to analgesic request | 24 hours
  Time to analgesic request
Quality of life (QoL) after laparoscopic cholecystectomy (LC) | 3 months
  Gastrointestinal Quality of Life Index questionnaire for QOL assessment with calculation of the score; most desirable option: 4 points, least desirable option: 0 points and GIQLI score: sum of the point. GIQLI ranges from 0 to 80 with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hepatology and Tropical Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No